CLINICAL TRIAL: NCT06203626
Title: Ultra-Low Field (ULF) Point Of Care (POC) MRI System for Study Brain Morphology and Pathology
Brief Title: Ultra-Low Field (ULF) Point-of-Care (POC) MRI System for Brain Morphology and Pathology
Status: Recruiting | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10001719; 001719-N
Record Dates: First submitted 2024-01-10; First posted 2024-01-12 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12-15

CONDITIONS: Nervous System Diseases (C10 Unique ID D009422)
Keywords: MRI; Brain; Morphometry; ultra-low field MRI; Lesion
MeSH Terms: conditions — Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- participant: we will collect an ULF-MRI from all participants.

SUMMARY:
Background:

Magnetic resonance imaging (MRI) is a tool for getting pictures of the tissues and organs inside the body. MRI can help diagnose many injuries and diseases. But not all patients are equally likely to receive MRIs. Factors such as race or ethnicity, distance to imaging centers, mobility, and a lower income can limit some people s access to MRIs. A new ultra-low field (ULF) type of MRI, which can be used on a vehicle, may help take imaging scans to more people. But researchers need to know that UFL-MRI works just as well as standard MRIs.

Objective:

To learn whether UFL-MRI is as good as standard MRI at detecting neurological disorders.

Eligibility:

People aged 3 years or older who have or show symptoms of neurological disease (such as stroke, cancer, or epilepsy). Healthy adults are also needed.

Design:

Participants will have 1 or 2 study visits.

Adult participants will have a physical exam. They will receive two MRI exams:

* Standard MRI. They will lie still on a narrow bed that will move into a large tube. They will wear earplugs to muffle the sounds.
* ULF-MRI. They will lie on a stretcher, and only their head will be inside a smaller tube. The noises will be quieter. They will wear earplugs to muffle the sounds.

Some adults may receive a contrast agent given through a small tube attached to a needle in the arm. The contrast agent helps the researchers see differences in the body more clearly. This may be done during 1 or both MRIs.

Children will have only 1 ULF-MRI.

Some participants may be invited to have additional visits for up to 6 months.

DETAILED DESCRIPTION:
Study Description:

Within the long-term goal of establishing a mobile research unit, this protocol aims at better understanding the utility and applicability of ULF MRI to deliver accessible neuroimages that could provide an opportunity for increasing participation in research, for early therapeutic intervention, and for potentially improvement of standard of care. For this purpose, we will invite healthy volunteers and populations with neurological presentations, mostly those enrolled in NIH studies collecting standard brain MRI, to participate in this protocol for ULF-MRI data collection. We will evaluate ULF MRI images in comparison to the standard field images. This analysis will aid at defining the type of research we can do with the ULF as a stand-alone technique and provide preliminary data for future research.

Based on the different clinical presentations, ancillary measures, such as cognitive, motor, and fatigue scales, optical coherence tomography, fundus, or blood samples, among others, might be collected to provide guidance for future studies.

Objectives:

Primary Objectives:

* Measure the ULF-MRI sensitivity to detect presence of pathology using the standard field MRI as the gold standard.
* To provide a framework for technical development.

Secondary Objective:

Describe participants social determinants of health.

Endpoints:

Primary Endpoint: ULF-MRI sensitivity to detect presence of pathology in comparison to the standard field MRI measured in 100 cases.

Secondary Endpoints: Descriptive participation.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Volunteer of any gender, 3 years of age and older.
* Adult participant: must be capable of understanding the procedures and requirements of this study and be able and willing to sign an informed consent document.
* Minor participant: Must have a parent or guardian capable of understanding the procedures and requirements of this study who are willing to sign an informed parental consent document, and where feasible, the minor age 7 and older provides assent.
* Either:

  * Adult in good general health as evidenced by medical history or
  * Diagnosed with a stroke, a neurological or neuro-oncological disease, or
  * Exhibiting symptoms suggestive of neurological or neuro-oncological disease.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Unable to undergo MRI study based on screening (e.g., presence of non-MRI compatible objects).
* Pregnancy or lactation, if contrast agent is required.

Ages: 3 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Healthy volunteers, Patients with previously identified brain anomalies, Patients with known or suspected neurological or neuro-oncological disorders, Stroke patients.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-03-26 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
ULF-MRI sensitivity to detect presence of pathology | Visit 1 and optional visit two within 180 days.
  ULF-MRI sensitivity to detect presence of pathology in comparison to the standard field MRI measured in 100 cases. A study will be considered to have a positive finding if the clinical report from the MRI brain collected at standard field has an observation.
Technical development | Visit 1 and optional repeated visits through the life of the protocol.
  Optimization of acquisition parameters, reproducibility, and training of personnel.

SECONDARY OUTCOMES:
Social determinants of health among participants | Visit 1.
  Characterizing the distribution of participants in our neuroimaging study.

CONTACTS AND LOCATIONS:
Overall Officials: Silvina G Horovitz, Ph.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
ULF MRI images with collaborators; ULF-MRI, standard MRI, other data upon tech transfer agreement; IPD that is required for publications.
Supporting Information: Study Protocol, Analytic Code
Time Frame: ULF-MRI with collaborator upon data collection upon request and agreement as required by publications.
Access Criteria: images and other relevant IPD information can be shared upon agreement. PI will review requests.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001719-N.html